CLINICAL TRIAL: NCT04470947
Title: Comprehensive Genomic Profiling and Next Generation Functional Drug Screening for Patients With Aggressive Haematological Malignancies: Next Generation Personal Hematology
Brief Title: Comprehensive Genomic Profiling and Next Generation Functional Drug Screening for Patients With Aggressive Haematological Malignancies
Acronym: EXALT-2
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Roche Pharma AG (Industry); Allcyte GmbH (Unknown)
Responsible Party: Principal Investigator, Philipp Staber, MD, PhD, Assoc. Prof. Priv.-Doz. Dr.med.univ. Philipp Staber, Medical University of Vienna
Other Study IDs: FA711C1050
Record Dates: First submitted 2020-07-07; First posted 2020-07-14 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Advanced Lymphoma; Refractory Lymphoma; Refractory Leukemia; Refractory Acute Myeloid Leukemia; Refractory T-Cell Lymphoma
Keywords: Personalized medicine
MeSH Terms: conditions — Lymphoma; Leukemia; Leukemia, Myeloid, Acute; Lymphoma, T-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Next generation functional drug screening
  Interventions: Diagnostic Test: Next generation functional drug screening; Diagnostic Test: Comprehensive genomic profiling
- Comprehensive genomic profiling
  Interventions: Diagnostic Test: Next generation functional drug screening; Diagnostic Test: Comprehensive genomic profiling
- Physician's choice
  Interventions: Diagnostic Test: Next generation functional drug screening; Diagnostic Test: Comprehensive genomic profiling

INTERVENTIONS:
Diagnostic Test: Next generation functional drug screening — High-throughput image based in-vitro drug screening on primary patient tumor cells
Diagnostic Test: Comprehensive genomic profiling — Comprehensive targeted profiling of genetic aberrations on primary patient tumor material
  Other Names: FoundationOne Heme

SUMMARY:
EXALT-2 is a prospective, randomized, three arm study for treatment decision guided either by either comprehensive genomic profiling, next generation drug screening or physician's choice

ELIGIBILITY:
Inclusion Criteria:

* patient is suffering from aggressive haematological disease AND has undergone at least two lines of previous therapies AND/OR has undergone at least one previous therapy and no standard treatment is available in the specific disease setting and disease specific guidelines recommend treatment in studies.
* duration of last response is less than 6 months defined as first day of last treatment to date of relapse, the response duration has to be available with dates (dd/mm/yyyy) for initiation of and relapse to previous treatment.
* best response to previous treatment has to be available.
* The patient is able to give written informed consent and wishes to undergo further therapy
* further therapy is medically feasible
* tumor cell-containing samples can be obtained

Exclusion Criteria:

* current participation in another experimental clinical trial
* performance status does not allow participation (ECOG ˃ 1)
* pregnancy, tested at screening
* patient suffers from classical or nodular, lymphocyte predominant Hodgkins lymphoma.
* other malignoma, diagnosed <1a before inclusion (except localized squamous cell carcinoma of the skin, surgically curable melanoma of the skin, basal cell carcinoma of the skin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 patients with relapsed/ refractory acute leukemia and relapsed/ refractory aggressive lymphoma after standard treatment fulfilling inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-06-10 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with a ratio ≥1.3 of progression free survival (PFS) compared to most recent treatment | Through study completion, an average of 8 month
  The study aims to identify if next-generation functional drug screening (ngFDS) and/or comprehensive genomic profiling (CGP; FoundationOne®Heme) compared to physicians' choice guided treatment will have an increased percentage of patients with a ratio
  ≥1.3 of progression free survival (PFS)/PFS of most recent treatment in patients with aggressive haematological malignancies

SECONDARY OUTCOMES:
Average Ratio of PFS/PFS of most prior treatment | Through study completion, an average of 8 months
  Average Ratio of PFS/PFS of most prior treatment
Overall response rate (ORR) | Through study completion, an average of 8 months
  Overall response rate (ORR)
Number of treatable targets identified | Through study completion, an average of 8 months
  Number of treatable targets identified

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Snijder B, Vladimer GI, Krall N, Miura K, Schmolke AS, Kornauth C, Lopez de la Fuente O, Choi HS, van der Kouwe E, Gultekin S, Kazianka L, Bigenzahn JW, Hoermann G, Prutsch N, Merkel O, Ringler A, Sabler M, Jeryczynski G, Mayerhoefer ME, Simonitsch-Klupp I, Ocko K, Felberbauer F, Mullauer L, Prager GW, Korkmaz B, Kenner L, Sperr WR, Kralovics R, Gisslinger H, Valent P, Kubicek S, Jager U, Staber PB, Superti-Furga G. Image-based ex-vivo drug screening for patients with aggressive haematological malignancies: interim results from a single-arm, open-label, pilot study. Lancet Haematol. 2017 Dec;4(12):e595-e606. doi: 10.1016/S2352-3026(17)30208-9. Epub 2017 Nov 15. PMID 29153976